CLINICAL TRIAL: NCT01506895
Title: A Phase 2, Multi-national, Multi-centre, Double Masked, Randomised, Placebo Controlled, Parallel-group Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Darapladib Administered for 3 Months to Adult Subjects With Diabetic Macular Edema With Centre Involvement
Brief Title: A Phase 2 Clinical Study to Investigate Effects of Darapladib in Subjects With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 115403
Record Dates: First submitted 2011-12-21; First posted 2012-01-10 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Retinopathy, Diabetic
Keywords: Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- darapladib (Experimental): darapladib dosed at 160 mg once daily
  Interventions: Drug: darapladib
- placebo (Placebo Comparator): Placebo to match once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: darapladib — Experimental compound 160 mg dose
  Arms: darapladib
Drug: placebo — Placebo to match
  Arms: placebo

SUMMARY:
The purpose of this study is to characterize the systemic and ocular safety and tolerability, pharmacokinetics, exploratory efficacy and pharmacodynamics of 3 months of repeat administration of oral darapladib in diabetic macular edema patients with centre involvement.

DETAILED DESCRIPTION:
This is a multi-national, multi-centre, randomised, double-masked, placebo-controlled, parallel-group study of repeat oral administration of 160 mg darapladib for 3 months in adult subjects with DME with centre involvement.

Eligible subjects will be randomised in a 2:1 ratio of active treatment to placebo, with the placebo group to allow a comparison of safety between treatment arms and to minimize the open label effect that can be observed with the visual acuity endpoint.

The primary aim of the study is to determine the effect of repeat doses of darapladib on the mean change from baseline of both best-corrected visual acuity (BCVA) and spectral domain OCT (SD-OCT) centre subfield. The study eye will be examined for changes over the life of the study. As this investigational treatment is systemic, the fellow eye may be examined in tandem to provide additional data.

ELIGIBILITY:
Inclusion Criteria:

* A female subject is eligible to participate if she is of: Non-childbearing potential or child-bearing potential and agrees to contraception for an appropriate period of time
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Confirmation of DME in the study eye by angiography
* Confirmation of retinal thickening in the study eye by study doctor
* Best corrected visual acuity score of 78-24 letters in the study eye

Exclusion Criteria:

* Additional eye disease in the study eye that could compromise study assessments
* Intraocular surgery, or laser photocoagulation in the study eye within 3 months of dosing
* Uncontrolled intraocular pressure in the study eye despite treatment with glaucoma medication
* Uncontrolled diabetes
* Certain types of liver disease
* Severe reduction in kidney function OR removal of a kidney OR kidney transplant
* Blood pressure higher than normal despite lifestyle changes and treatment with medications
* Certain medications that may interfere with the study medication or eye assessments (these will be identified by the study doctor)
* Current severe heart failure
* Severe asthma that is poorly controlled with medication
* Previous severe allergic reaction to food, medications, drink, insect stings, etc
* If both birth parents are at least 50% Japanese, Chinese, or Korean ancestry, must have a blood sample collected for Lp-PLA2 activity. Those with Lp-PLA2 activity less than or equal to 20.0 nmol/min/mL are excluded
* Recent participation in a study of an investigational medication
* Any other reason the investigator deems the subject should not participate in the study
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Visual Acuity as measured by ETDRS BCVA | 3 months
  Mean change from baseline in ETDRS Best Corrected Visual Acuity (BCVA) after 3 months of treatment
Change from baseline in Spectral Domain Optical Coherance Tomography | 3 months
  Mean change from baseline in SD-OCT after 3 months of treatment

SECONDARY OUTCOMES:
Changes in Retinal Anatomy | 3 months
  Changes in retinal anatomy as assessed by fluorescein angiography and fundus photography and SD-OCT in the study eye
Safety and Tolerability as assessed by change from baseline in outcome measures | 3 months
  Safety and tolerability as assesed by: change from baseline in blood pressure and heart rate; assessed by change from baseline in complete ophthalmic exam and visual acuity; assessed by change from baseline in clinical laboratory tests; assessed by change from baseline in the collection of adverse events
Changes in Pharmacodynamic LP-PLA2 enzyme inhibition | 3 months
  Changes over 3 months in the study of LP-PLA2 Enzyme inhibition as data permit
Peak plasma concentration (Cmax) of study drug | 3 months
  Plasma Pharmacokinetic parameters of darapladib as data permit
Plasma concentration versus time curve (AUC) of study drug | 3 months
  Plasma Pharmacokinetic parameters of darapladib as data permit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Australia (4):
  - GSK Investigational Site, Parramatta, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- GSK Investigational Site, Glostrup Municipality, Denmark
- Germany (5):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
- Italy (3):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Padua, Veneto
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115403 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register